CLINICAL TRIAL: NCT00622700
Title: An International, Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Two Year Treatment With Teriflunomide 7 mg Once Daily and 14 mg Once Daily Versus Placebo in Patients With a First Clinical Episode Suggestive of Multiple Sclerosis Plus a Long Term Extension Period
Brief Title: Phase III Study With Teriflunomide Versus Placebo in Patients With First Clinical Symptom of Multiple Sclerosis
Acronym: TOPIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6260; HMR1726D-3005 (Other: HMR); 2006-001152-12 (EudraCT Number)
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Multiple Sclerosis
Keywords: MS; Clinically Isolated Syndrome; CIS; CDMS; relapses
MeSH Terms: conditions — Multiple Sclerosis; Recurrence | interventions — teriflunomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo/Teriflunomide 7 mg or Teriflunomide 14 mg (Placebo Comparator): Core treatment period: Placebo matched to teriflunomide tablet once daily orally.
  Extension treatment period: Re-randomized in 1:1 ratio to either teriflunomide 7 mg or 14 mg once daily orally.
  Interventions: Drug: Teriflunomide; Drug: Placebo
- Teriflunomide 7 mg/7 mg (Experimental): Core treatment period: Teriflunomide 7 mg tablet once daily orally.
  Extension treatment period: Teriflunomide 7 mg tablet once daily orally.
  Interventions: Drug: Teriflunomide
- Teriflunomide 14 mg/14 mg (Experimental): Core treatment period: Teriflunomide 14 mg tablet once daily orally.
  Extension treatment period: Teriflunomide 14 mg tablet once daily orally.
  Interventions: Drug: Teriflunomide

INTERVENTIONS:
Drug: Teriflunomide — Film-coated tablet Oral administration
  Other Names: HMR1726; Aubagio
Drug: Placebo — Film-coated tablet Oral administration
  Arms: Placebo/Teriflunomide 7 mg or Teriflunomide 14 mg

SUMMARY:
The primary objective was to demonstrate the effect of teriflunomide (HMR1726) (14 milligram per day [mg/day] and 7 mg/day), in comparison to placebo, for reducing conversion of participants presenting with their first clinical episode consistent with multiple sclerosis (MS) to clinically definite multiple sclerosis (CDMS).

The secondary objectives were:

* To demonstrate the effect of teriflunomide, in comparison to placebo, on:

  * Reducing conversion to definite multiple sclerosis (DMS)
  * Reducing annualized relapse rate (ARR)
  * Reducing disease activity/progression as measured by Magnetic Resonance Imaging (MRI)
  * Reducing accumulation of disability for at least 12 weeks as measured by the Expanded Disability Status Scale (EDSS)
  * Proportion of disability-free participants as assessed by the EDSS
  * Reducing participant-reported fatigue
* To evaluate the safety and tolerability of teriflunomide
* To evaluate the pharmacokinetics (PK) of teriflunomide
* Optional pharmacogenomic testing aimed at assessing the association between the main enzyme systems of teriflunomide metabolism and hepatic safety, and other potential associations between gene variations and clinical outcomes

DETAILED DESCRIPTION:
The study consisted of 4 periods:

* Screening period: up to 4 weeks,
* Placebo-controlled treatment period: up to 108 weeks (at least 24 weeks for participants who experienced conversion to CDMS),
* Extension treatment period (without placebo-control): the extension period continued until teriflunomide was commercially available in participant's country of residence.
* Post-treatment washout period: 4 weeks after last treatment intake.

The maximal duration of the study period per participant was expected to be 116 weeks if he/she did not continue in the extension treatment period.

ELIGIBILITY:
Inclusion Criteria:

* First acute or subacute, well-defined neurological event consistent with demyelination (that is, optic neuritis confirmed by an ophthalmologist, spinal cord syndrome, brainstem/cerebellar syndromes)
* Onset of MS symptoms occurring within 90 days of randomization
* A screening MRI scan with 2 or more T2 lesions at least 3 millimeter (mm) in diameter that are characteristic of MS

Exclusion Criteria:

* Clinically relevant cardiovascular, hepatic, neurological, endocrine or other major systemic disease
* Significantly impaired bone marrow function
* Pregnancy or nursing
* Alcohol or drug abuse
* Use of cladribine, mitoxantrone, or other immunosuppressant agents such as azathioprine, cyclophosphamide, cyclosporin, methotrexate or mycophenolate before enrollment
* Any known condition or circumstance that would prevent in the investigator's opinion compliance or completion of the study

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 618 (Actual)
Dates: Start 2008-02; Primary Completion 2012-12 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (131):
- United States (19):
  - Investigational Site Number 8965, Cullman, Alabama
  - Investigational Site Number 8954, Phoenix, Arizona
  - Investigational Site Number 8946, Phoenix, Arizona
  - Investigational Site Number 8962, Fort Collins, Colorado
  - Investigational Site Number 8920, Maitland, Florida
  - Investigational Site Number 8953, St. Petersburg, Florida
  - Investigational Site Number 8914, Fort Wayne, Indiana
  - Investigational Site Number 8940, Indianapolis, Indiana
  - Investigational Site Number 8922, Shreveport, Louisiana
  - Investigational Site Number 8955, Grand Rapids, Michigan
  - Investigational Site Number 8949, Traverse City, Michigan
  - Investigational Site Number 8937, St Louis, Missouri
  - Investigational Site Number 8951, Albuquerque, New Mexico
  - Investigational Site Number 8925, New York, New York
  - Investigational Site Number 8941, Charlotte, North Carolina
  - Investigational Site Number 8924, Dayton, Ohio
  - Investigational Site Number 8905, Round Rock, Tennessee
  - Investigational Site Number 8930, Burlington, Vermont
  - Investigational Site Number 8963, Seattle, Washington
- Australia (4):
  - Investigational Site Number 1405, Geelong
  - Investigational Site Number 1404, Heidelberg
  - Investigational Site Number 1407, Hobart
  - Investigational Site Number 1401, Parkville
- Austria (3):
  - Investigational Site Number 4004, Innsbruck
  - Investigational Site Number 4005, Linz
  - Investigational Site Number 4001, Vienna
- Bulgaria (6):
  - Investigational Site Number 5312, Pleven
  - Investigational Site Number 5307, Sofia
  - Investigational Site Number 5304, Sofia
  - Investigational Site Number 5309, Sofia
  - Investigational Site Number 5303, Sofia
  - Investigational Site Number 5306, Sofia
- Canada (8):
  - Investigational Site Number 5402, Greenfield Park
  - Investigational Site Number 5403, London
  - Investigational Site Number 5409, Montreal
  - Investigational Site Number 5401, Ottawa
  - Investigational Site Number 5406, Québec
  - Investigational Site Number 5408, Sherbrooke
  - Investigational Site Number 5410, Toronto
  - Investigational Site Number 5404, Toronto
- Chile (4):
  - Investigational Site Number 5602, Santiago
  - Investigational Site Number 5601, Santiago
  - Investigational Site Number 5606, Santiago
  - Investigational Site Number 5605, Viña del Mar
- Czechia (4):
  - Investigational Site Number 5801, Brno
  - Investigational Site Number 5803, Hradec Králové
  - Investigational Site Number 5804, Olomouc
  - Investigational Site Number 5805, Ostrava - Poruba
- Denmark (2):
  - Investigational Site Number 6002, Aarhus C
  - Investigational Site Number 6004, Esbjerg
- Estonia (2):
  - Investigational Site Number 6201, Tallinn
  - Investigational Site Number 6203, Tartu
- Finland (3):
  - Investigational Site Number 6405, Helsinki
  - Investigational Site Number 6403, Kuopio
  - Investigational Site Number 6401, Turku
- France (9):
  - Investigational Site Number 6611, Besançon
  - Investigational Site Number 6601, Clermont-Ferrand
  - Investigational Site Number 6609, Lille
  - Investigational Site Number 6604, Montpellier
  - Investigational Site Number 6612, Nancy
  - Investigational Site Number 6605, Nantes
  - Investigational Site Number 6602, Nice
  - Investigational Site Number 6614, Nîmes
  - Investigational Site Number 6607, Strasbourg
- Germany (10):
  - Investigational Site Number 6801, Bayreuth
  - Investigational Site Number 6810, Berlin
  - Investigational Site Number 6805, Berlin
  - Investigational Site Number 6807, Erbach im Odenwald
  - Investigational Site Number 6803, Essen
  - Investigational Site Number 6809, Hanover
  - Investigational Site Number 6804, Ludwigshafen
  - Investigational Site Number 6815, Minden
  - Investigational Site Number 6802, Münster
  - Investigational Site Number 6806, Wiesbaden
- Hungary (4):
  - Investigational Site Number 7101, Budapest
  - Investigational Site Number 7103, Budapest
  - Investigational Site Number 7108, Esztergom
  - Investigational Site Number 7105, Veszprém
- Lithuania (3):
  - Investigational Site Number 7402, Klaipėda
  - Investigational Site Number 7403, Šiauliai
  - Investigational Site Number 7401, Vilnius
- Mexico (2):
  - Investigational Site Number 7501, Chihuahua City
  - Investigational Site Number 7502, Guadalajara
- Poland (5):
  - Investigational Site Number 7709, Gdansk
  - Investigational Site Number 7710, Lodz
  - Investigational Site Number 7701, Warsaw
  - Investigational Site Number 7703, Warsaw
  - Investigational Site Number 7707, Warsaw
- Romania (5):
  - Investigational Site Number 7803, Bucharest
  - Investigational Site Number 7806, Bucharest
  - Investigational Site Number 7805, Cluj-Napoca
  - Investigational Site Number 7807, Cluj-Napoca
  - Investigational Site Number 7808, Timișoara
- Russia (8):
  - Investigational Site Number 7907, Kazan'
  - Investigational Site Number 7909, Nizhny Novgorod
  - Investigational Site Number 7906, Nizhny Novgorod
  - Investigational Site Number 7904, Nizhny Novgorod
  - Investigational Site Number 7912, Novosibirsk
  - Investigational Site Number 7910, Rostov-on-Don
  - Investigational Site Number 7911, Saint Petersburg
  - Investigational Site Number 7905, Smolensk
- Turkey (Türkiye) (11):
  - Investigational Site Number 8304, Edirne
  - Investigational Site Number 8309, Istanbul
  - Investigational Site Number 8315, Istanbul
  - Investigational Site Number 8308, Istanbul
  - Investigational Site Number 8310, Istanbul
  - Investigational Site Number 8312, Istanbul
  - Investigational Site Number 8305, Izmir
  - Investigational Site Number 8301, Izmir
  - Investigational Site Number 8303, Izmir
  - Investigational Site Number 8302, İzmit
  - Investigational Site Number 8314, Trabzon
- Ukraine (11):
  - Investigational Site Number 8507, Chernihiv
  - Investigational Site Number 8501, Dnipropetrovsk
  - Investigational Site Number 8511, Donets'K
  - Investigational Site Number 8506, Kharkiv
  - Investigational Site Number 8504, Kharkiv
  - Investigational Site Number 8508, Kiev
  - Investigational Site Number 8512, Lutsk
  - Investigational Site Number 8505, Lviv
  - Investigational Site Number 8510, Poltava
  - Investigational Site Number 8503, Vinnytsia
  - Investigational Site Number 8502, Zaporizhzhya
- United Kingdom (8):
  - Investigational Site Number 8709, Liverpool
  - Investigational Site Number 8701, London
  - Investigational Site Number 8704, London
  - Investigational Site Number 8706, Newcastle upon Tyne
  - Investigational Site Number 8705, Nottingham
  - Investigational Site Number 8708, Plymouth
  - Investigational Site Number 8707, Salford
  - Investigational Site Number 8702, Sheffield

REFERENCES:
- [Background] Miller AE, Wolinsky JS, Kappos L, Comi G, Freedman MS, Olsson TP, Bauer D, Benamor M, Truffinet P, O'Connor PW; TOPIC Study Group. Oral teriflunomide for patients with a first clinical episode suggestive of multiple sclerosis (TOPIC): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Neurol. 2014 Oct;13(10):977-86. doi: 10.1016/S1474-4422(14)70191-7. Epub 2014 Sep 2. PMID 25192851

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 846 participants were screened, of which 618 randomized in core treatment period. Out of 618, 423 entered in extension treatment period. End date of core treatment period was 17 December 2012 (maximum treatment duration: 120 weeks). End date of extension treatment period was 05 February 2016 (maximum treatment duration: 283 weeks).
Pre-assignment Details: Participants were randomized in 1:1:1 ratio to teriflunomide 7 mg,14 mg or placebo in core treatment period. Those completing core period, given opportunity to enter long-term extension period (participants originally given placebo re-randomized [1:1]to teriflunomide 7 mg/14 mg; those originally given 7 mg,14 mg continued with the same fixed dose).
Groups:
- Placebo: Core treatment period: Placebo matched to teriflunomide tablet once daily orally.
- Teriflunomide 7 mg: Core treatment period: Teriflunomide 7 mg tablet once daily orally.
- Teriflunomide 14 mg: Core treatment period: Teriflunomide 14 mg tablet once daily orally.
- Placebo/ Teriflunomide 7 mg: Core treatment period: Placebo matched to teriflunomide tablet once daily orally.
  Extension treatment period: Teriflunomide 7 mg tablet once daily orally.
- Placebo/Teriflunomide 14 mg: Core treatment period: Placebo matched to teriflunomide tablet once daily orally.
  Extension treatment period: Teriflunomide 14 mg tablet once daily orally.
Period: Core Treatment Period
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg | Placebo/ Teriflunomide 7 mg | Teriflunomide 7 mg/7 mg | Placebo/Teriflunomide 14 mg | Teriflunomide 14 mg/14 mg
Started | 197 | 205 | 216 | 0 | 0 | 0 | 0
Treated | 197 | 203 | 214 | 0 | 0 | 0 | 0
Completed | 141 | 150 | 163 | 0 | 0 | 0 | 0
Not Completed | 56 | 55 | 53 | 0 | 0 | 0 | 0
Not completed — Randomized but Not Treated | 0 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 18 | 25 | 18 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 19 | 6 | 12 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 3 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 18 | 15 | 0 | 0 | 0 | 0
Not completed — Other than specified above | 2 | 2 | 5 | 0 | 0 | 0 | 0
Period: Extension Treatment Period
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg | Placebo/ Teriflunomide 7 mg | Teriflunomide 7 mg/7 mg | Placebo/Teriflunomide 14 mg | Teriflunomide 14 mg/14 mg
Started | 0 (Participants were re-randomized in a 1:1 ratio to either teriflunomide 7 mg or 14 mg treatment arm.) | 0 | 0 | 64 (10 participants completed core treatment period but did not enter in extension treatment period.) | 142 (8 participants completed core treatment period but did not enter in extension treatment period.) | 67 (10 participants completed core treatment period but did not enter in extension treatment period.) | 150 (13 participants completed core treatment period but did not enter in extension treatment period.)
Completed | 0 | 0 | 0 | 43 | 103 | 50 | 120
Not Completed | 0 | 0 | 0 | 21 | 39 | 17 | 30
Not completed — Adverse Event | 0 | 0 | 0 | 5 | 9 | 6 | 8
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 8 | 1 | 9
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 1 | 2 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 11 | 16 | 6 | 10
Not completed — Missing | 0 | 0 | 0 | 2 | 3 | 1 | 0
Not completed — Other than specified above | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized population: all randomized participants according to the treatment group to which they were assigned in the core treatment period.
Groups:
- Placebo: Placebo matched to teriflunomide tablet once daily orally.
- Teriflunomide 7 mg: Teriflunomide 7 mg tablet once daily orally.
- Teriflunomide 14 mg: Teriflunomide 14 mg tablet once daily orally.
- Total: Total of all reporting groups
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg | Total
Number analyzed (Participants) | 197 | 205 | 216 | 618
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (8.4) | 31.6 (9.0) | 32.8 (8.1) | 32.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 130 | 154 | 419
  Male | 62 | 75 | 62 | 199
Region [Number; unit: participants]
  Eastern Europe | 94 | 96 | 101 | 291
  Western Europe | 76 | 74 | 74 | 224
  Americas and Australia | 27 | 35 | 41 | 103
Expanded Disability Status Scale (EDSS) Score [Mean (Standard Deviation); unit: units on a scale] — EDSS is an ordinal scale in half-point increments that qualifies disability in participants with MS. It consists of 8 ordinal rating scales assessing seven functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS).
  units on a scale | 1.71 (1.00) | 1.50 (1.02) | 1.80 (0.97) | 1.67 (1.00)

OUTCOME MEASURES:

1. Primary Outcome: Core Treatment Period: Time to Conversion to Clinically Deﬁnite Multiple Sclerosis (CDMS)
Description: Conversion to CDMS was defined by the occurrence of a relapse, which was defined as a new neurological abnormality separated by at least 30 days from onset of a preceding clinical event, presented for at least 24 hours and occurred in the absence of fever or known infection. Percent probability of conversion at 24, 48, and 108 weeks was estimated using Kaplan-Meier method.
Time Frame: Up to a maximum of 108 weeks depending on time of enrollment
Population: Intent-to-treat (ITT) population included all randomized participants who had at least 1 day study medication exposure. Participants were analyzed in the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 197 | 203 | 214
percent probability
  Percent Probability of Conversion at 24 weeks | 14.3 [9.2 to 19.4] | 8.7 [4.6 to 12.8] | 9.0 [5.0 to 13.0]
  Percent Probability of Conversion at 48 weeks | 26.0 [19.2 to 32.8] | 14.2 [8.9 to 19.6] | 13.7 [8.6 to 18.7]
  Percent Probability of Conversion at 108 weeks | 35.9 [27.8 to 43.9] | 27.6 [19.9 to 35.4] | 24.0 [17.0 to 31.0]
Statistical Analysis 1: Comparison: Placebo vs Teriflunomide 14 mg; A step-down hierarchical testing procedure, starting with the test of teriflunomide 14 mg versus placebo was used. Time to conversion to CDMS was analyzed using the Cox proportional hazard model with treatment, region, and baseline monofocal/multifocal status as covariates; Test type: Superiority or Other; p = 0.0087, Wald chi-squared — P value was derived using Wald chi-squared test in the Cox proportional hazard model; Hazard Ratio (HR) = 0.574, 95% CI 2-sided [0.379 to 0.869]
Statistical Analysis 2: Comparison: Placebo vs Teriflunomide 7 mg; A step-down hierarchical testing procedure was used. The second step was the test of teriflunomide 7 mg versus placebo for time to conversion to CDMS. Time to conversion to CDMS was analyzed using the Cox proportional hazard model with treatment, region, and baseline monofocal/multifocal status as covariates; Test type: Superiority or Other; p = 0.0271, Wald chi-squared — P value was derived using Wald chi-squared test in the Cox proportional hazard model; Hazard Ratio (HR) = 0.628, 95% CI 2-sided [0.416 to 0.949]

2. Secondary Outcome: Core Treatment Period: Time to Conversion to Definite Multiple Sclerosis (DMS)
Description: Conversion to DMS was demonstrated by dissemination of MRI lesions in time (as per McDonald criteria) or a relapse, whichever occurs first. MRI Imaging criteria were detection of Gadolinium (Gd) enhancement at least 3 months after onset of initial clinical event, if not at site corresponding to initial event; detection of new T2 lesion if it appears at any time compared with reference scan (done at time of screening) done at least 30 days after onset of the initial clinical event. Occurrence of relapse was defined as new neurological abnormality separated by at least 30 days from onset of preceding clinical event, present for at least 24 hours and occurring in absence of fever or known infection. New clinical abnormality (neurological sign) that is consistent with participant's symptoms with increase in at least one Functional System (FS) or EDSS score compared to last EDSS assessment. Percent probability of conversion at 24, 48, and 108 weeks was estimated using Kaplan-Meier method.
Time Frame: Up to a maximum of 108 weeks depending on time of enrollment
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 197 | 203 | 214
percent probability
  Percent Probability of Conversion at 24 weeks | 58.2 [51.0 to 65.4] | 45.7 [38.5 to 52.9] | 46.0 [39.0 to 53.0]
  Percent Probability of Conversion at 48 weeks | 72.4 [65.7 to 79.1] | 57.3 [49.8 to 64.7] | 57.8 [50.6 to 64.9]
  Percent Probability of Conversion at 108 weeks | 87.0 [81.2 to 92.7] | 73.3 [66.0 to 80.7] | 71.5 [64.5 to 78.4]
Statistical Analysis 1: Comparison: Placebo vs Teriflunomide 14 mg; A step-down hierarchical testing procedure was used. The third step was the test of teriflunomide 14 mg versus placebo for time to conversion to DMS. This was analyzed using the Cox proportional hazard model with treatment, region, and baseline monofocal/multifocal status as covariates; Test type: Superiority or Other; p = 0.0003, Wald chi-squared — P value was derived using Wald chi-squared test in the Cox proportional hazard model; Hazard Ratio (HR) = 0.651, 95% CI 2-sided [0.515 to 0.822]
Statistical Analysis 2: Comparison: Placebo vs Teriflunomide 7 mg; A step-down hierarchical testing procedure was used. The fourth step was the test of teriflunomide 7 mg versus placebo for time to conversion to DMS. This was analyzed using the Cox proportional hazard model with treatment, region, and baseline monofocal/multifocal status as covariates; Test type: Superiority or Other; p = 0.0020, Wald chi-squared — P value was derived using Wald chi-squared test in the Cox proportional hazard model; Hazard Ratio (HR) = 0.686, 95% CI 2-sided [0.540 to 0.871]

3. Secondary Outcome: Core Treatment Period: Annualized Relapse Rate (ARR)
Description: ARR is the total number of confirmed relapses that occurred during the treatment period divided by the total number of patient-years treated. Each episode of relapse (appearance, or worsening of a clinical symptom that was stable for at least 30 days, that persisted for a minimum of 24 hours in the absence of fever) was to be confirmed by an increase in EDSS score or Functional System scores. ARR was assessed using Poisson regression model with robust error variance. To account for the different treatment durations among participants, a Poisson regression model with robust error variance was used (total number of confirmed relapses onset between randomization date and last dose date as the response variable, treatment, region and baseline monofocal/multifocal status as covariates, and log-transformed treatment duration as an offset variable).
Time Frame: Up to a maximum of 108 weeks depending on time of enrollment
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: relapses per patient year
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 197 | 203 | 214
relapses per patient year | 0.284 [0.214 to 0.378] | 0.190 [0.139 to 0.260] | 0.194 [0.143 to 0.263]

4. Secondary Outcome: Core Treatment Period: Brain Magnetic Resonance Imaging (MRI) Assessment: Change From Baseline in Total Lesion Volume at Week 108
Description: The total lesion volume (burden of disease) is the total volumes of hyperintense on T2 plus hypointense on T1 as measured by MRI scan. Least-square means were estimated using a Mixed-effect model with repeated measures (MMRM) on cubic root transformed volume data with factors for treatment, baseline monofocal/multifocal status, region, visit, treatment-by-visit interaction, cubic root transformed baseline burden of disease, and baseline-by-visit interaction.
Time Frame: Baseline, Week 108
Population: ITT population, but including only participants who had post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: milliliter
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 68 | 75 | 99
milliliter | 0.053 (0.033) | 0.041 (0.032) | -0.038 (0.029)

5. Secondary Outcome: Core Treatment Period: Brain MRI Assessment: Number of Gadolinium Enhancing (Gd-enhancing) T1-lesions Per MRI Scan (Poisson Regression Estimates)
Description: Number of Gd-enhancing T1-lesions per scan is the total number of Gd-enhancing T1-lesions that occurred during the treatment period divided by the total number of scans performed during the treatment period. To account for the different numbers of scans performed among the participants, a Poisson regression model with robust error variance was used (total number of Gd-enhancing T1-lesions as response variable, treatment, baseline monofocal/multifocal status, region and baseline number of Gd-enhancing T1-lesions as covariates, and log-transformed number of scans as an offset variable).
Time Frame: Up to a maximum of 108 weeks depending on time of enrollment
Population: ITT population, but including only participants who had post-baseline data.
Measure: Number (95% Confidence Interval); unit: lesions per scan
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 109 | 84 | 74
lesions per scan | 0.953 [0.708 to 1.284] | 0.749 [0.433 to 1.294] | 0.395 [0.262 to 0.598]

6. Secondary Outcome: Core Treatment Period: Brain MRI Assessment: Volume of Gadolinium Enhancing (Gd-enhancing) T1-lesions Per MRI Scan
Description: Total volume of Gd-enhancing T1-lesions per scan is the sum of the volumes of Gd-enhancing T1-lesions observed during the treatment period divided by the total number of scans performed during the treatment period. To account for the different numbers of scans performed among the participants, a Poisson regression model with robust error variance was used (total number of Gd-enhancing T1-lesions as response variable, treatment, baseline monofocal/multifocal status, region and baseline number of Gd-enhancing T1-lesions as covariates, and log-transformed number of scans as an offset variable).
Time Frame: Up to a maximum of 108 weeks depending on time of enrollment
Population: ITT population, but including only participants who had post-baseline data.
Measure: Number; unit: milliliters per scan
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 109 | 84 | 74
milliliters per scan | 0.079 | 0.058 | 0.034

7. Secondary Outcome: Core Treatment Period: Brain MRI Assessment: Change From Baseline in Volume of Hypointense Post-Gadolinium T1 Lesion Component
Description: Volume of hypointense post-gadolinium T1 lesion component was measured by MRI scan. Least-square means were estimated using a Mixed-effect model with repeated measures (MMRM) on cubic root transformed volume data adjusted for baseline monofocal/multifocal status, region, visit, treatment-by-visit interaction, cubic root transformed baseline value, and baseline-by-visit interaction
Time Frame: Baseline, Week 108
Population: ITT population, but including only participants who had post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: milliliter
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 68 | 75 | 99
milliliter | 0.028 (0.018) | 0.025 (0.018) | -0.033 (0.016)

8. Secondary Outcome: Core Treatment Period: Brain MRI Assessment: Change From Baseline in Volume of T2 Lesion Component
Description: Volume of T2 lesion component was measured by MRI scan. Least-square means were estimated using a Mixed-effect model with repeated measures (MMRM) on cubic root transformed volume data adjusted for baseline monofocal/multifocal status, region, visit, treatment-by-visit interaction, cubic root transformed baseline value, and baseline-by-visit interaction.
Time Frame: Baseline, Week 108
Population: ITT population, but including only participants who had post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: milliliter
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 68 | 75 | 99
milliliter | 0.052 (0.033) | 0.036 (0.032) | -0.035 (0.029)

9. Secondary Outcome: Core Treatment Period: Brain MRI Assessment: Percent Change From Baseline in Atrophy
Description: Atrophy was measured by MRI scan.
Time Frame: Baseline, Week 108
Population: ITT population, but including only participants who had post-baseline data.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 68 | 75 | 99
percent change | -0.386 (1.326) | -0.197 (1.218) | -0.366 (1.151)

10. Secondary Outcome: Core Treatment Period: Time to 12-Week Sustained Disability Progression
Description: The 12-week sustained disability progression was defined as increase from baseline of at least 1-point in EDSS score (at least 0.5-point for participants with baseline EDSS score of greater than [>] 5.5) that persisted for at least 12 weeks. Percent probability of participants free of 12-week sustained disability progression at 24, 48, and 108 weeks was estimated using Kaplan-Meier method.
Time Frame: Up to a maximum of 108 weeks depending on time of enrollment
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 197 | 203 | 214
percent probability
  Percent Probability at 24 weeks | 96.0 [93.0 to 98.9] | 94.3 [90.9 to 97.8] | 97.9 [95.9 to 99.9]
  Percent Probability at 48 weeks | 91.7 [87.3 to 96.1] | 90.1 [85.4 to 94.7] | 93.9 [90.2 to 97.6]
  Percent Probability at 108 weeks | 85.5 [79.2 to 91.8] | 86.5 [80.8 to 92.1] | 89.2 [84.1 to 94.3]

11. Secondary Outcome: Core Treatment Period: Change From Baseline in EDSS at Week 108
Description: EDSS is an ordinal scale in half-point increments that qualifies disability in participants with MS. It consists of 8 ordinal rating scales assessing seven functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS). Least-square means were estimated using a Mixed-effect model with repeated measures (MMRM) on cubic root transformed volume data adjusted for baseline monofocal/multifocal status, region, visit, treatment-by-visit interaction, baseline value and baseline-by-visit interaction
Time Frame: Baseline, Week 108
Population: ITT population, but including only participants who had post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 80 | 82 | 102
units on a scale | 0.069 (0.087) | -0.191 (0.086) | -0.166 (0.080)

12. Secondary Outcome: Core Treatment Period: Change From Baseline in Fatigue Impact Scale (FIS) Total Score at Week 108
Description: FIS is a participant-reported scale that qualifies the impact of fatigue on daily life in participants with MS. It consists of 40 statements that measure fatigue in three areas; physical, cognitive, and social. FIS total score ranges from 0 (no problem) to 160 (extreme problem). Least-square means were estimated using a Mixed-effect model with repeated measures [MMRM] on FIS total score data adjusted for or baseline monofocal/multifocal status, region, visit, treatment-by-visit interaction, baseline value and baseline-by-visit interaction.
Time Frame: Baseline, Week 108
Population: ITT population, but including only participants who had post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 84 | 95 | 106
units on a scale | -2.537 (2.794) | -2.524 (2.710) | -1.827 (2.551)

13. Secondary Outcome: Core Treatment Period: Overview of Adverse Events (AEs)
Description: AEs are any unfavorable and unintended sign, symptom, syndrome, or illness observed by the investigator or reported by the participant during the study.
Time Frame: From first study drug intake up to 112 days after last intake in the placebo-controlled period or up to first intake in the extension treatment period, whichever occurred first
Population: Safety population:all randomized participants exposed to study medication; analyzed according to drug actually received. In Placebo arm, 4 received teriflunomide 7mg & 2 received teriflunomide 14mg, hence they were included in respective teriflunomide arm. Participants who were randomized but not treated were excluded (2 in each teriflunomide arm).
Measure: Number; unit: participants
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 191 | 207 | 216
participants
  Any AE | 155 | 161 | 183
  Any serious AE | 18 | 18 | 24
  Any AE leading to death | 1 | 0 | 0
  Any AE leading to treatment discontinuation | 19 | 25 | 18

14. Secondary Outcome: Extension Treatment Period: Time to Conversion to Clinically Deﬁnite Multiple Sclerosis (CDMS)
Description: Conversion to CDMS was defined by the occurrence of a relapse, which was defined as a new neurological abnormality separated by at least 30 days from onset of a preceding clinical event, presented for at least 24 hours and occurred in the absence of fever or known infection. Percent probability of conversion was estimated using Kaplan-Meier method.
Time Frame: From randomization in the core period up to 390 Weeks (Extension treatment period [maximum exposure: 283 Weeks])
Population: ITT Population: all randomized participants in the extension who had at least 1 day IMP exposure. Participants were analyzed according to the treatment group allocated by the randomization in the core study followed by the re-randomized treatment group during the extension period.
Measure: Number (95% Confidence Interval); unit: Percent probability
Groups:
- Placebo/Teriflunomide 7 mg; Teriflunomide 7 mg/ 7mg: Core treatment period: Placebo matched to teriflunomide tablet once daily orally.
  Extension treatment period: Teriflunomide 7 mg tablet once daily orally.
- Placebo/ Teriflunomide 14 mg: Core treatment period: Placebo matched to teriflunomide tablet once daily orally.
  Extension treatment period: Teriflunomide 14 mg tablet once daily orally.
Arm/Group | Placebo/Teriflunomide 7 mg | Teriflunomide 7 mg/ 7mg | Placebo/ Teriflunomide 14 mg | Teriflunomide 14 mg/14 mg
Number analyzed (Participants) | 64 | 142 | 67 | 150
Percent probability
  Percent Probability of Conversion at 24 Weeks | 4.7 [0.0 to 9.9] | 3.5 [0.5 to 6.6] | 13.5 [5.3 to 21.6] | 4.7 [1.3 to 8.0]
  Percent Probability of Conversion at 48 Weeks | 12.5 [4.4 to 20.6] | 9.9 [5.0 to 14.8] | 21.2 [11.3 to 31.0] | 8.7 [4.2 to 13.3]
  Percent Probability of Conversion at 72 Weeks | 15.7 [6.8 to 24.6] | 17.1 [10.9 to 23.4] | 24.3 [13.9 to 34.6] | 14.8 [9.1 to 20.6]
  Percent Probability of Conversion at 96 Weeks | 18.9 [9.3 to 28.6] | 23.9 [16.7 to 31.0] | 27.4 [16.6 to 38.2] | 16.2 [10.3 to 22.1]
  Percent Probability of Conversion at 120 Weeks | 22.3 [12.0 to 32.7] | 27.7 [20.2 to 35.2] | 32.2 [20.8 to 43.6] | 18.3 [12.1 to 24.6]
  Percent Probability of Conversion at 144 Weeks | 22.3 [12.0 to 32.7] | 29.4 [21.7 to 37.1] | 33.9 [22.3 to 45.4] | 22.0 [15.3 to 28.8]
  Percent Probability of Conversion at 168 Weeks | 22.3 [12.0 to 32.7] | 32.2 [24.2 to 40.3] | 33.9 [22.3 to 45.4] | 22.8 [16.0 to 29.7]
  Percent Probability of Conversion at 192 Weeks | 22.3 [12.0 to 32.7] | 37.5 [28.6 to 46.4] | 35.9 [24.0 to 47.8] | 24.8 [17.6 to 32.0]
  Percent Probability of Conversion at 216 Weeks | 25.6 [13.9 to 37.3] | 38.9 [29.8 to 48.1] | 39.3 [26.3 to 52.3] | 24.8 [17.6 to 32.0]
  Percent Probability of Conversion at 240 Weeks | 29.5 [16.1 to 42.9] | 40.8 [31.3 to 50.4] | 39.3 [26.3 to 52.3] | 26.3 [18.7 to 34.0]
  Percent Probability of Conversion at 264 Weeks | 29.5 [16.1 to 42.9] | 43.0 [32.9 to 53.2] | 39.3 [26.3 to 52.3] | 26.3 [18.7 to 34.0]
  Percent Probability of Conversion at 288 Weeks | 29.5 [16.1 to 42.9] | 43.0 [32.9 to 53.2] | 39.3 [26.3 to 52.3] | 26.3 [18.7 to 34.0]
  Percent Probability of Conversion at 312 Weeks | 29.5 [16.1 to 42.9] | 43.0 [32.9 to 53.2] | 49.4 [28.3 to 70.5] | 26.3 [18.7 to 34.0]
  Percent Probability of Conversion at 336 Weeks | 29.5 [16.1 to 42.9] | 48.7 [34.7 to 62.7] | 49.4 [28.3 to 70.5] | 26.3 [18.7 to 34.0]

15. Secondary Outcome: Extension Treatment Period: Overview of Adverse Events (AEs)
Description: AEs are any unfavorable and unintended sign, symptom, syndrome, or illness observed by the investigator or reported by the participant during the study. Safety population included all randomized population who actually received at least 1 dose of the IMP in extension and analyzed according to the treatment actually received in core study followed by treatment actually received in the extension treatment period.
Time Frame: From re-randomization up to 283 Weeks
Population: Analysis was performed on Safety population. In Placebo/teriflunomide 7mg arm, 2 received 7mg in the core period; In Placebo/teriflunomide 14mg, 1 received 7mg in the core period, hence, they were included in the 7mg/7mg arm in extension period as treatment received in the core period for consistency.
Measure: Number; unit: participants
Groups:
- Teriflunomide 7 mg/ 7mg: Core treatment period: Teriflunomide 7 mg tablet once daily orally.
  Extension treatment period: Teriflunomide 7 mg tablet once daily orally.
Arm/Group | Placebo/Teriflunomide 7 mg | Teriflunomide 7 mg/ 7mg | Placebo/ Teriflunomide 14 mg | Teriflunomide 14 mg/14 mg
Number analyzed (Participants) | 62 | 145 | 66 | 150
participants
  Any AE | 47 | 110 | 57 | 120
  Any Serious AE | 8 | 17 | 8 | 24
  Any AE Leading to Death | 0 | 0 | 0 | 0
  Any AE leading to Permanent Discontinuation | 5 | 8 | 5 | 7

16. Other Pre Specified Outcome: Core Treatment Period: Liver Function: Number of Participants With Potentially Clinically Significant Abnormalities (PCSA)
Description: PCSA values are abnormal values considered medically important by the Sponsor according to predefined criteria based on literature review.
  Hepatic parameters thresholds were defined as follows:
  * Alanine Aminotransferase (ALT) >3, 5, 10 or 20 upper limit of normal(ULN);
  * Aspartate aminotransferase (AST) >3, 5, 10 or 20 ULN;
  * Alkaline Phosphatase >1.5 ULN;
  * Total Bilirubin (TB) >1.5, 2, or 3 ULN;
  * ALT >3 ULN and TB >2 ULN.
Time Frame: as for outcome 13
Population: Safety population as described in Outcome Measure 13. Here 'n' signifies the number of participants for the treatment group who had that parameter assessed at post-baseline.
Measure: Number; unit: participants
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 191 | 207 | 216
participants
  ALT >3 ULN (n=190, 207, 216) | 18 | 25 | 26
  ALT >5 ULN (n=190, 207, 216) | 12 | 10 | 11
  ALT >10 ULN (n=190, 207, 216) | 5 | 1 | 3
  ALT >20 ULN (n=190, 207, 216) | 0 | 0 | 1
  AST >3 ULN (n=190, 207, 216) | 9 | 12 | 10
  AST >5 ULN (n=190, 207, 216) | 1 | 4 | 6
  AST >10 ULN (n=190, 207, 216) | 1 | 0 | 1
  AST >20 ULN (n=190, 207, 216) | 0 | 0 | 1
  Alkaline Phosphatase >1.5 ULN (n=190, 207, 216) | 0 | 0 | 1
  TB >1.5 ULN (n=190, 207, 216) | 14 | 9 | 8
  TB >2 ULN (n=190, 207, 216) | 8 | 0 | 3
  TB >3 ULN (n=190, 207, 216) | 0 | 0 | 1
  ALT >3 ULN and TB >2 ULN (n=190, 207, 216) | 2 | 0 | 2

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (up to 390 weeks [maximum exposure in core treatment period: 120 weeks and maximum exposure in extension treatment period: 283 weeks]) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from first dose of study drug up to 112 days after last intake in core treatment period [or up to 1st intake in extension period, whichever occurred first] or 28 days after last intake in extension treatment period). Analysis was performed on safety population as described in Outcome Measure 15.
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg | Placebo/Teriflunomide 7 mg | Teriflunomide 7 mg/7 mg | Placebo/Teriflunomide 14 mg | Teriflunomide 14 mg/14 mg
Serious Adverse Events (participants affected / at risk) | 18/191 | 18/207 | 24/216 | 8/62 | 17/145 | 8/66 | 24/150
Other Adverse Events (participants affected / at risk) | 117/191 | 129/207 | 135/216 | 33/62 | 66/145 | 38/66 | 70/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=191) | Teriflunomide 7 mg (N=207) | Teriflunomide 14 mg (N=216) | Placebo/Teriflunomide 7 mg (N=62) | Teriflunomide 7 mg/7 mg (N=145) | Placebo/Teriflunomide 14 mg (N=66) | Teriflunomide 14 mg/14 mg (N=150)
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Genital infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 2 | 1 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psychiatric decompensation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radicular syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Axonal neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dental cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Radicular cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 0 | 1 | 1 | 0
Cervical cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fallopian tube cyst (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Testicular torsion (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hernia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 2 | 0 | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 5 | 4 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=191) | Teriflunomide 7 mg (N=207) | Teriflunomide 14 mg (N=216) | Placebo/Teriflunomide 7 mg (N=62) | Teriflunomide 7 mg/7 mg (N=145) | Placebo/Teriflunomide 14 mg (N=66) | Teriflunomide 14 mg/14 mg (N=150)
Nasopharyngitis (Infections and infestations) | 29 | 24 | 35 | 9 | 14 | 9 | 15
Bronchitis (Infections and infestations) | 5 | 9 | 8 | 4 | 7 | 2 | 8
Sinusitis (Infections and infestations) | 9 | 7 | 6 | 6 | 4 | 4 | 6
Influenza (Infections and infestations) | 9 | 8 | 16 | 3 | 5 | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 14 | 23 | 20 | 2 | 5 | 2 | 4
Urinary tract infection (Infections and infestations) | 10 | 10 | 20 | 3 | 5 | 5 | 4
Depression (Psychiatric disorders) | 11 | 8 | 8 | 2 | 4 | 3 | 1
Headache (Nervous system disorders) | 25 | 31 | 30 | 4 | 8 | 8 | 6
Dizziness (Nervous system disorders) | 7 | 7 | 11 | 1 | 4 | 2 | 4
Paraesthesia (Nervous system disorders) | 9 | 11 | 22 | 3 | 1 | 3 | 4
Hypertension (Vascular disorders) | 2 | 5 | 12 | 3 | 4 | 0 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 11 | 2 | 0 | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 22 | 15 | 4 | 9 | 4 | 14
Nausea (Gastrointestinal disorders) | 9 | 11 | 9 | 2 | 7 | 1 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 12 | 25 | 2 | 3 | 7 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 14 | 8 | 4 | 5 | 4 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 13 | 7 | 1 | 4 | 2 | 4
Fatigue (General disorders) | 14 | 10 | 9 | 2 | 3 | 4 | 3
Alanine aminotransferase increased (Investigations) | 28 | 32 | 35 | 0 | 5 | 6 | 3
Blood creatine phosphokinase increased (Investigations) | 1 | 9 | 5 | 4 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.